CLINICAL TRIAL: NCT06644235
Title: The Impact of Cold Application on Pain and Comfort During the Process of Diabetic Foot Care
Brief Title: Pain and Comfort in Diabetic Foot Ulcer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, HEDİYE UTLİ, Assistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/109-4
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus
Keywords: diabetic foot ulser; pain; cold application; comfort
MeSH Terms: conditions — Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cold Application Group (Experimental): Measurements were taken from the participants in the intervention group in DFU care before (sociodemographic data, the Site, Ischemia, Neuropathy, Bacterial Infection, and Depth (SINBAD) score, score, HbA1c level, pain and comfort levels), during (pain) and after (pain and comfort) cold application.
  Interventions: Other: Cold Application
- Control Group (No Intervention): The solution was used at room temperature (+18°C to +24°C) as used in routine care without any intervention in DFU care.

INTERVENTIONS:
Other: Cold Application — Before DFU care, the patient was given an appropriate position and the materials (forceps, scalpel, sponge, pad, bandage, etc.) and the temperature of the 0.9% NaCl solution kept in the refrigerator for 24 hours were measured with an infrared thermometer (+4°C to +8°C) and taken to the treatment area. The solution was transferred to a 50 mL syringe in a sterile manner. The solution was instilled into the wound simultaneously with wound care (5-15 min).
  Arms: Cold Application Group

SUMMARY:
The purpose of this study is to reveal the effect of cold application of 0.9% NaCl solution used during diabetic foot ulcer (DFU) care on the pain and comfort levels of patients. In this direction; - Cold application has no effect on pain and comfort levels in DFU care. - Cold application has an effect on pain and comfort levels in DFU care. Hypotheses were created. In order to reveal the effect of cold application, 0.9% NaCl was compared to the intervention group (+4ͦ C and +8ͦ C); NaCl ( sodium chloride) compared to the control group (+18ͦ C and +24ͦ C).

DETAILED DESCRIPTION:
Diabetic foot ulcer (DFU) prevalence is increasing in parallel with the increasing number of patients with diabetes mellitus (DM). Patients experience pain due to debridement, which is frequently used in DFU care. Therefore, it is seen that nonpharmacological strategies are needed in pain management, unlike pharmacological methods. For this purpose, this single-blind randomized controlled study attempted to provide more information to the literature for supportive care in DFU care. 68 DFU patients were included in the study. After being randomly assigned to the groups, the care solution was applied cold or hot according to the procedure in the DFU care performed in the outpatient clinic. Data were collected before (10 min before), during and after (10 min after) the procedure. Kruskal Wallis, One Way ANOVA, Post Hoc pairwise comparison tests and corrected Bonferroni were used in the analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 with a diabetic foot wound diagnosed with diabetes mellitus,
* No cognitive impairment,
* No hearing, understanding or speaking problems,
* VAS>3 points,
* Patients who consent to participate in the study

Exclusion Criteria:

* Patients who have been decided to have an intervention to reduce pain before the procedure (such as local anesthesia, nerve blockade, opioid analgesics, etc.) -Patients with VAS <3 points,
* Patients with arterial or venous ulcers other than DFU

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Pain | 45 minutes (Time to collect data from each patient)
  Pain level was expressed through VAS pain scale; value of "0 = no pain", "1-3 = mild pain", "4-6 = moderate pain", "7-9 = severe pain" and "10 = unbearable pain". While evaluating the pain, the patient marked the facial expression corresponding to his pain.
Comfort | 45 minutes (Time to collect data from each patient)
  Comfort was measured using the General Comfort Scale Short Form (GCS-SF). The 28-item six-point Likert scale is scored between 28 and 168. It is accepted that the comfort level increases as the score increases.

SECONDARY OUTCOMES:
SINBAD score | 45 minutes (Time to collect data from each patient)
  The diabetic foot wound assessment (SINBAD) score is a scoring system that evaluates diabetic wounds in 6 categories (1. zone; 2. ischemia, 3. neuropathy, 4. bacterial infection, 5. ulcer area, 6. depth). It is an easy, fast and simple classification that is used by giving 0 or 1 points to each category, with a maximum of 6 points.

CONTACTS AND LOCATIONS:
Overall Officials: Mensure Turan, PhD, Principal Investigator — Şırnak Üniversitesi
Locations (1):
- Health Sciences University Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No